CLINICAL TRIAL: NCT06797518
Title: A Multicenter, Single Arm, Open Label Biopsy Study to Evaluate Structural and Functional Changes in Kidneys of Adult Patients With IgA Nephropathy Receiving Iptacopan on Top of Supportive Care
Brief Title: Study to Evaluate the Impact of Iptacopan on Top of SOC on Biopsy Changes in Kidneys of Adult Patients With IgAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023A2201
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Glomerulonephritis, IGA; Immunoglobulin A Nephropathy
Keywords: IgAN, Renal Biopsy, Iptacopan
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — iptacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Iptacopan (Experimental): All the study participants will receive iptacopan 200 mg oral capsule b.i.d, while remaining on the maximally tolerated or locally approved maximal daily doses of ACEi/ARB throughout the treatment period.
  Interventions: Drug: Iptacopan

INTERVENTIONS:
Drug: Iptacopan — LNP023 oral capsule 200 mg b.i.d
  Other Names: LNP023

SUMMARY:
A study to investigate the impact of iptacopan treatment on the underlying immunopathology in patients with IgAN by assessing changes in key clinical and molecular markers from baseline to 9 months. The study aims to provide insights into the treatment's systemic and kidney-specific aspects by quantifying the change in mesangial C3c containing fragments deposition, as an indicator of complement activation, and evaluating a variety of biomarkers related to kidney function, damage, and disease progression, including but not limited to Oxford MEST-C score.

DETAILED DESCRIPTION:
The study comprises of a screening period followed by a baseline visit, at which a baseline kidney biopsy will be performed. Eligible participants included in the study will receive iptacopan 200 mg b.i.d for a 9-month treatment period. Dose adjustment of iptacopan is not allowed during the treatment period. At Month 9, upon completion of the treatment period, a follow up biopsy is performed for all participants at the time of end of study (EOS).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study; participants should be able to communicate well with the investigator, understand and comply with the requirements of the study.
2. Male and female participants ≥18 years of age with biopsy-confirmed IgA nephropathy and an eGFR ≥ 30 mL/min/1.73m2. eGFR will be calculated using the CKD-EPI 2009 formula.
3. Proteinuria as assessed at screening by UPCR ≥ 0.8g/g or 1g/d sampled from FMV.
4. Biopsy at baseline should confirm IgAN with < 50% tubulointerstitial fibrosis.
5. Participants must be on ACEi or ARB treatment at either the locally approved maximal daily dose or the maximally tolerated dose (per investigators' judgment) for approximately 90 days prior to baseline visit and continue on a stable dose throughout the study. Participants with allergies or intolerance to ACEi and ARB are eligible for the study, but the investigator should clearly document the reasons for not being on maximal ACEi/ARB dose in the source documents. In addition, if participants are taking diuretics, other antihypertensive medication or Sodium-Glucose Co-Transporter 2 inhibitors (SGLT2i), the doses should be stabilized for at least 90 days prior to baseline.
6. Vaccination against Neisseria meningitidis and Streptococcus pneumoniae infections required to be completed at least 2 weeks prior to the start of study treatment. If the participants have not been previously vaccinated, or if a booster is required, vaccine should be given according to local regulations at least 2 weeks prior to first study drug administration. If study treatment must start earlier than 2 weeks post-vaccination, prophylactic antibiotic treatment should be initiated.
7. Vaccination against Haemophilus influenzae infection should be given, if available and according to local regulations, at least 2 weeks prior to first study drug administration.

Exclusion Criteria:

1. Any secondary IgAN (at historic or baseline biopsies) as defined by the investigator and IgA vasculitis Henoch-Scholein Purpura (HSP). Secondary IgAN can be associated with cirrhosis, celiac disease, Human Immunodeficiency Virus (HIV) infection, dermatitis herpetiformis, seronegative arthritis, small-cell carcinoma, lymphoma, disseminated tuberculosis, bronchiolitis obliterans, and inflammatory bowel disease, familial Mediterranean fever, etc.
2. Any secondary diagnosis at baseline biopsy (other than IgA nephropathy).
3. Evidence of significant urinary obstruction or difficulty in voiding; any urinary tract disorder other than IgAN at screening and before first study drug administration.
4. Current or planned usage of any homeopathic and/or herbal medications for IgAN disease progression, such as but not limited to Lei Gong Teng.
5. Current acute kidney injury (AKI) defined by Acute Kidney Injury Network (AKIN) criteria within 4 weeks of screening.
6. Presence of rapidly progressive glomerulonephritis (RPGN) as defined by 50% decline in eGFR within 3 months prior to screening, or presence of nephrotic syndrome.
7. Sitting office SBP >140 mmHg or DBP >90 mmHg at the screening visit.
8. Participants treated with immunosuppressive or other immunomodulatory agents such as but not limited to cyclophosphamide, rituximab, infliximab, eculizumab, canakinumab, mycophenolate mofetil (MMF) or mycophenolate sodium (MPS), cyclosporine, tacrolimus, sirolimus, everolimus, systemic corticosteroids exposure (>7.5 mg/d prednisone/prednisolone equivalent) or targeted release formulation (TRF) of budesonide within 90 days (or 180 days for rituximab) prior to first study drug administration. Participants using other medication such us hydroxychloroquine or Endothelin receptor antagonists (ERAs).
9. Use of other investigational drugs within 5 half-lives or within 30 days of enrollment, whichever is longer.
10. Prior use of iptacopan or prior enrollment in any other iptacopan clinical trial where study drug was taken, including matching placebo.
11. All transplanted participants (any solid organ transplantation, including bone marrow transplantation).
12. History of recurrent invasive infections caused by encapsulated organisms, such as meningococcus and pneumococcus.
13. Major concurrent comorbidities including but not limited to advanced cardiac disease (e.g., New York Heart Association (NYHA) class IV), severe pulmonary disease (e.g., severe pulmonary hypertension (World Health Organization (WHO) class IV)), or hepatic disease (e.g., active hepatitis) that in the opinion of the investigator precludes participant's participation in the study.
14. Any medical condition deemed likely to interfere with the participant's participation in the study or that will require the use of prohibited medications.
15. Active systemic bacterial, viral (including COVID-19) or fungal infection within 14 days prior to study drug administration.
16. Presence of fever ≥ 38°C (100.4°F) within 7 days prior to study drug administration.
17. Human immunodeficiency virus (HIV) infection (known history of HIV or test positive for HIV antibody at Screening).
18. History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes.
19. Liver disease, such as active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection defined as positive HBsAg in conjunction with core antibody (anti-HBc), or HCV-RNA positive at screening, or liver injury as indicated by abnormal liver function tests at screening as defined below:

    * Any single parameter of ALT, AST, GGT, alkaline phosphatase must not exceed 3 × upper limit of normal (ULN)
    * Serum bilirubin must not exceed 2 × ULN
20. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer treated with curative intent), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
21. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (HCG) laboratory test.
22. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they agree to use effective methods of contraception during dosing of investigational drug and for 1 week after stopping of investigational drug.

Effective contraception methods include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks before taking investigational drug. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Male sterilization (at least 6 months prior to screening) of male partner of the female participant.
* Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps). For UK: with spermicidal foam/gel/film/cream/vaginal suppository.
* Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS).
* In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking investigational drug.
* If local regulations are more stringent than the contraception methods listed above, local regulations apply and will be described in the ICF.
* Women are considered post-menopausal if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms). Women are considered not of childbearing potential if they are post-menopausal or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential.
* If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the ICF.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-11-27 (Estimated); Study Completion 2027-11-27 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving a reduction of minimum one order of magnitude in complement C3c mesangial deposition. | BSL, Month 9
  Mesangial C3c deposition is assessed by intensity of immunofluorescence (IF) staining using the following grading system: 0 (absent) 1 (+) 2 (++) 3 (+++)

SECONDARY OUTCOMES:
Change from baseline at 9 months in CD68 cells | BSL, Month 9
  To describe the histopathological changes in additional biomarkers after treatment with iptacopan
Change from baseline at 9 months in staining of Immunoglobulins (IgA and IgG) | BSL, Month 9
  To describe the histopathological changes in additional biomarkers after treatment with iptacopan

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA Medical Center, Los Angeles, California
  - Nephronet Clinical, Buford, Georgia
  - CaRe Research, Chubbuck, Idaho
  - DaVita Clinical Research, Las Vegas, Nevada
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Prolato Clinical Research Center, Houston, Texas
- Novartis Investigative Site, CABA, Buenos Aires, Argentina
- Israel (4):
  - Novartis Investigative Site, Ashdod
  - Novartis Investigative Site, Hadera
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Nahariya
- Novartis Investigative Site, Kuala Lumpur, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com